CLINICAL TRIAL: NCT02466932
Title: Effects of Birth Weight on Anterior Eye Segment Measurements in Full-Term Children by Galilei Dual-Scheimpflug Analyzer
Status: Completed | Type: Observational
Sponsor: Neon Hospital (Other)
Collaborators: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Volkan YETER, Dr., Neon Hospital
Other Study IDs: 2010-171
Record Dates: First submitted 2015-06-03; First posted 2015-06-09 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Birth Weight
MeSH Terms: conditions — Birth Weight

STUDY DESIGN:
Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Birth Weight
  Interventions: Device: Galilei Dual-Scheimpflug Analyzer

INTERVENTIONS:
Device: Galilei Dual-Scheimpflug Analyzer — Measuring of Anterior Segment by Galilei Dual-Scheimpflug Analyzer

SUMMARY:
This study evaluates the effects of birth weight (BW) on ocular anterior segment parameters in preschool children using the Galilei Dual-Sheimpflug Analyzer (GD-SA). Children were measured by GD-SA and relationships between all anterior segment parameters obtained by this device and birth weight were analyzed.

DETAILED DESCRIPTION:
Preschoolers, who were born heavier, had thicker cornea and lens, longer axial length, and flatter corneal curve. The thicknesses and axial curves of central cornea within 7mm may be particularly associated with BW.

ELIGIBILITY:
Inclusion Criteria:

* ages 3- 6 years;
* birth weight >2,500 g;
* gestational age (i.e., the period of time between the first day of the mother's last menstrual period and birth) >37 weeks;
* visual acuity >0.8 (in decimals);
* no history of any systemic or ocular diseases;
* no history of previous ocular surgeries;
* no retinopathy of prematurity;
* no current medications; and
* no retinal or optic disc abnormalities on fundoscopy.

Exclusion Criteria:

* ages <3 >6 years;
* birth weight <2,500 g;
* gestational age (i.e., the period of time between the first day of the mother's last menstrual period and birth) <37 weeks;
* visual acuity <0.8 (in decimals);
* history of any systemic or ocular diseases;
* history of previous ocular surgeries;
* retinopathy of prematurity;
* current medications; and
* retinal or optic disc abnormalities on fundoscopy.

Ages: 30 Months to 80 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy children aged between 3-6- preschoolers- born at term and have birth weight heavier than 2500g
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2011-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Measurements of anterior segment parameters in Full-Term Children by Galilei Dual-Scheimpflug Analyzer | 1 day
  Corneal parameters, anterior chamber parameters and lens thickness were measured by Galilei Dual-Scheimpflug Analyzer in healthy preschool children.